CLINICAL TRIAL: NCT05110443
Title: A Comparison of Static and Dynamic PET/CT in Patients With Malignancies, Infections and Inflammatory Diseases (HYPOTHESIS Generation Study)
Brief Title: A Comparison of Static and Dynamic PET/CT (HYPOTHESIS Generation Study)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, André H. Dias, Principal Investigator, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYPOTHESIS
Record Dates: First submitted 2021-10-13; First posted 2021-11-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Oncology; Infections; Inflammation
Keywords: PET/CT; FDG; Dynamic Whole-Body
MeSH Terms: conditions — Neoplasms; Infections; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm (Other): Patients will perform a D-WB PET/CT scan as a substitute for their clinical PET.
  Interventions: Other: D-WB PET/CT

INTERVENTIONS:
Other: D-WB PET/CT — Instead of the usual procedure of having the injection of the radiotracer in the waiting room and having to wait 60 minutes before being moved to the scanner room for imaging, the study participants will be injected with the radiotracer already laying on the scanner bed and the scan will commence immediately.
  Therefore, in this study the patients are still only being scanned once, but we are gathering PET information in a different way.

SUMMARY:
The general purpose of this initial study is to evaluate whether parametric PET/CT improves diagnosis and treatment monitoring in select diseases. The specific aim of the HYPOTHESIS GENERATION study is:

1. To obtain and compare parametric as well as traditional static PET/CT images and determine the number of lesions identified on each type of scan.

DETAILED DESCRIPTION:
The hypothesis generating study will include a wide range of patients scheduled for PET/CT as part of either pre-therapy staging or treatment response.

Most scans will be performed with FDG, with indications for PET/CT including hematological, urogenital, thoracic and gynecological malignancies as well as patients with suspected infections and inflammation. We will also include patients referred for PET/CT using other radiotracers, such as tumour markers (68Ga-DOTATOC, 18F-FDOPA, 68Ga-PSMA, 18F-PSMA).

Instead of the usual procedure of having the injection of the radiotracer in the waiting room and having to wait 60 minutes before being moved to the scanner room for imaging, the study participants will be injected with the radiotracer already laying on the scanner bed and the scan will commence immediately.

Therefore, in this study the patients are still only being scanned once, but we are gathering PET information in a different way.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a planned clinical standard PET/CT as part of pre-therapeutic staging, response assessment scanning or evaluation of infection/inflammation.
* Good performance status, which permits patients to lay still in the scanner for ca. 70 min.

Exclusion Criteria:

* Age < 18 or > 85 years
* Patients that can not tolerate a PET scan (f.ex: claustrophobia).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Obtaining a database of parametric and traditional static PET/CT images for comparison of visual and semiquantitative evaluation | through study completion, average 1 year
  We will perform a correlation of the image derived from parametric PET/CT with those obtained from static PET/CT. This will allow us to evaluate if there are clinical advantages in regards to using parametric PET in clinical routine.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
According to local rules and GDRP it is not possible for study data to leave the facility.

REFERENCES:
- [Derived] Pedersen MA, Dias AH, Hjorthaug K, Gormsen LC, Fledelius J, Johnsson AL, Borgquist S, Tramm T, Munk OL, Vendelbo MH. Increased lesion detectability in patients with locally advanced breast cancer-A pilot study using dynamic whole-body [18F]FDG PET/CT. EJNMMI Res. 2024 Mar 25;14(1):31. doi: 10.1186/s13550-024-01096-4. PMID 38528239